CLINICAL TRIAL: NCT04483492
Title: Direct Effect of Caffeine on Diaphragmatic Muscles
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, H. Tolga Çelik, Principal Investigator, Hacettepe University
Other Study IDs: KA-20029
Record Dates: First submitted 2020-06-25; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Caffeine
MeSH Terms: interventions — caffeine citrate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: newborns under 32 weeks with respiratory support if they are decided to start caffeine treatment
  Interventions: Drug: Caffeine citrate

INTERVENTIONS:
Drug: Caffeine citrate — diaphragm contractility after administration

SUMMARY:
The mechanism of methylxanthines is thought to increase chemoreceptor responsiveness to CO2 in central nervous system. Besides, effect of methylxanthines on diaphragmatic contractility has also been found in experimental studies. A study of premature newborns has showed caffeine increase diaphragmatic activity and tidal volume. But, there is limited data about caffeine direct effect on diaphragma.

Objective: The investigators aimed to show the direct effect of caffeine on diphragmatic contractility.

Method: The babies under 32 weeks with respiratory support, are being enrolled in this study if caffeine treatment is decided to receive. Evaluation of muscle contraction is being made by ultrasound before and 30 minutes after caffeine loading dose. Right and left sides of diaphragm thickness are being measured by two clinicians on B mode ultrasound by anterior subcostal view. The velocity before and after caffeine administration will be calculated, dividing excursion frequency (parameter) for inspiratory time. Movement of the diaphragm at inspiratory and expiratory phases are also observed on M mode and the difference between the two phases are measured.

ELIGIBILITY:
Inclusion Criteria:

* newborns under 32 weeks with respiratory support
* caffeine is decided to give

Exclusion Criteria:

* babies with congenital malformations

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: newborns under 32 weeks with respiratory support on their first week
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
diphragmatic contractility | 30 minutes
  diphragmatic contractility measured by ultrasonographic evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kraaijenga JV, Hutten GJ, de Jongh FH, van Kaam AH. The Effect of Caffeine on Diaphragmatic Activity and Tidal Volume in Preterm Infants. J Pediatr. 2015 Jul;167(1):70-5. doi: 10.1016/j.jpeds.2015.04.040. Epub 2015 May 15. PMID 25982138
- [Derived] Kayki G, Celik HT, Ayaz E, Tandircioglu UA, Oguz B, Yigit S, Yurdakok M. Direct Effect of Caffeine on Diaphragmatic Muscles in Preterm Babies Through Ultrasonographic Examination. Turk Arch Pediatr. 2024 Apr 5;59(3):277-282. doi: 10.5152/TurkArchPediatr.2024.23290. PMID 39140727